CLINICAL TRIAL: NCT02384018
Title: A Phase I Study Evaluating Safety and Tolerability of Autologous Bone Marrow-derived Mesenchymal Stromal Cells in Chronic Pancreatitis Patients Who Undergo Total Pancreatectomy and Islet Autotransplantation.
Brief Title: Mesenchymal Stem Cell and Islet Co-transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Hongjun Wang, Professor of Surgery, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CCT-BMMSC15-001; 5R21DK099696 (NIH)
Record Dates: First submitted 2014-12-16; First posted 2015-03-10 (Estimated); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Chronic Pancreatitis; Diabetes
MeSH Terms: conditions — Pancreatitis, Chronic; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Patients will receive standard islet transplantation.
- autologous mesenchymal stromal cell (Experimental): Patients will receive MSCs together with standard islet transplantation.
  Interventions: Biological: autologous mesenchymal stromal cell

INTERVENTIONS:
Biological: autologous mesenchymal stromal cell — Islet transplantation patients will receive autologous MSCs following islets infusion
  Arms: autologous mesenchymal stromal cell

SUMMARY:
The purpose of this study is to show safety and tolerability to our mesenchymal stromal cells (MSCs) product which will be autologous in nature, expanded using a non-xenogeneic, human component expansion media (pooled human platelet lysate) and delivered fresh. Subsequently, the investigators intend to test whether infusion of MSCs immediately after islet autograft can reduce onset of diabetes and improve glycemic control after total pancreatectomy and islet autotransplantation.

DETAILED DESCRIPTION:
This is a Phase I study evaluating safety and tolerability of autologous BM-MSCs in chronic pancreatitis patients who undergo total pancreatectomy and islet autotransplantation (TP-IAT). CCT-BMMSC will be infused at one of the following doses: (Tier 1), 20x10^6 cell per patient, (Tier 2), 50x10^6 cell per patient, and (Tier 3), 100x10^6 cell per patient.

Primary objective: To describe and compare the safety and tolerability of infusion of fresh autologous bone marrow-derived Mesenchymal stromal cells after islet transplantation in chronic pancreatitis patients who undergo TP-IAT. The investigators plan to enroll 24 patients for the whole study. The duration of this study is 12 months. The investigators anticipate that this study will be completed within 2 years of commencement.

Secondary objective: Efficacy of infusion of fresh autologous bone marrow-derived Mesenchymal stromal cells together after islet transplantation in chronic pancreatitis patients who undergo TP-IAT as assessed through onset of diabetes, glycemic control, pain relief and quality of life index.

Safety variables: Adverse events (AEs), Laboratory parameters (hematology, biochemistry, urinalysis), Vital signs

ELIGIBILITY:
Inclusion Criteria:

* Chronic pancreatitis patients who undergo TP-IAT.
* >18 years of age.
* Patients with BMI from 18.5 to 30.
* Renal function: >90mls/min/1.73m squared
* Normal INR/PT/PTT values for MUSC clinical laboratory standards
* Diabetes free before surgery (fasting blood glucose<125mg/dl).
* No prior pancreatic surgery with the exception of transduodenal sphincteroplasty or Whipple/Beger procedure.
* Patients with normal liver function as measured by serum levels of aminotransferase including alanine aminotransferase (ALT), and aspartate aminotransferase (AST), and total bilirubin levels.

Exclusion Criteria:

* Patients whose Hemoglobin, Hematocrit, and Platelet count are above or below normal values for MUSC clinical laboratory standards.
* Patients who has hematological malignancy.
* Patients who are under immunosuppression.
* Patients with marked calcification disease on CT scan.
* Patients with severe fibrosis and atrophy on pancreas MRI.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2017-11-21 (Actual)

PRIMARY OUTCOMES:
C-peptide level after mixed meal tolerance test | 12 months

SECONDARY OUTCOMES:
Liver function, kidney function | 12 months after transplant
The absence of severe hypoglycemic episodes | 12 months after transplant

CONTACTS AND LOCATIONS:
Overall Officials: Hongjun Wang, Ph.D, Principal Investigator — Medical University of South Carolina
Locations (1):
- GI Surgery, Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Result] Wang H, Strange C, Nietert PJ, Wang J, Turnbull TL, Cloud C, Owczarski S, Shuford B, Duke T, Gilkeson G, Luttrell L, Hermayer K, Fernandes J, Adams DB, Morgan KA. Autologous Mesenchymal Stem Cell and Islet Cotransplantation: Safety and Efficacy. Stem Cells Transl Med. 2018 Jan;7(1):11-19. doi: 10.1002/sctm.17-0139. Epub 2017 Nov 21. PMID 29159905